CLINICAL TRIAL: NCT04290585
Title: Text for Health: Integrating Technology and Health Communication to Improve Health Outcomes (Part 2 of 2)
Brief Title: Technology and Health Communication in Improving Health Outcomes in Patients Scheduled for Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB13858; NCI-2015-02088 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB13858 (Other: Fox Chase Cancer Center); P30CA006927 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Female Breast Carcinoma; Healthy Subject

ARMS (1):
- Health Services Research (text message reminder) (Experimental): Patients receive 1-2 text messages a few weeks before and 1 text message 24 hours before their mammography screening appointment. Patients also receive a phone call reminder as per standard practice.
  Interventions: Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive text message reminders

SUMMARY:
This pilot clinical trial studies how well technology and health communication works in improving health outcomes in patients scheduled for mammography screening. The Mobile Mammography Screening Program provides a vital health service and it is important that all women scheduled for an appointment show-up to be screened. Technology and health communication may help decrease no-show rates among patients scheduled for mammography screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To decrease the mobile mammography unit no-show rate by sending text message appointment reminders to patients.

II. To assess the efficacy of the text message reminders at addressing the no-show rate by collecting satisfaction survey data from patients that received the texts and that came to their scheduled appointment.

OUTLINE:

Patients receive 1-2 text messages a few weeks before and 1 text message 24 hours before their mammography screening appointment. Patients also receive a phone call reminder as per standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Appointment is at a participating location
* Has a cell phone that can send and receive text messages
* Agrees to receive the text messages
* Can read either English or Spanish
* Not yet sent text messages to 100 patients in community or corporate sites
* Scheduled at least 1 week prior to the appointment date
* PATIENTS FOR FOLLOW UP: come to their scheduled appointment
* PATIENTS FOR FOLLOW UP: received the text message reminders
* PATIENTS FOR FOLLOW UP: can read either English or Spanish

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2014-10-28 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in no-show rate pre- and post-intervention | Baseline to up to 1 year
  The change (or lack of change) in the corporate sites? no-show rate will be compared to the change (or lack of change) in the community sites? no-show rate. Descriptive statistics will be used to describe the results.

SECONDARY OUTCOMES:
Acceptability of using text messaging as a reminder: survey | Up to 1 year
  Descriptive statistics will be used to report the results of the satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Esnaola, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States